CLINICAL TRIAL: NCT06478745
Title: Trajectories and Experiences of Patients With Multimorbidity in the National Health Service of Spain: a Mixed Methods Study (LOXO-MULTIPAP)
Brief Title: Trajectories and Experiences of People With Multimorbidity in Spain (LOXO-MULTIPAP) Project: a Mixed Methods Study
Acronym: LOXO
Status: Enrolling by invitation | Type: Observational
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: PI. Bernardino Oliva. Instituto Investigación Sanitaria Illes Balears (Unknown); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); PI Antonio Gimeno. Instituto de Investigación Sanitaria Aragón. (Unknown); PI. Rafael Rotaeche. Instituto Investigación Bioguipuzcoa. Osakidetza (Unknown); PI. Francisca Leiva. Instituto de Investigacion Biomedica de Malaga. (Unknown); CI. Julian Librero. Navarra Biomed. Servicio Navarro de Salud (Unknown); Fundación Investigacion en Innovacion Biomédica en Atención Primaria FIIBAP (Unknown); Instituto de Investigación Sanitaria Gregorio Marañón (Other)
Responsible Party: Principal Investigator, Isabel Del Cura-Gonzalez, Principal - Coordinator researcher, Gerencia de Atención Primaria, Madrid
Other Study IDs: 20230033; PI22/00768 Isabel del Cura (Other Grant/Funding Number: Instituto Salud Carlos III-European Regional Develop. Found); PI22/01651 Francisca Leiva (Other Grant/Funding Number: Instituto Salud Carlos III-European Regional Development F.); PI22/00701 Antonio Gimeno (Other Grant/Funding Number: Instituto Salud Carlos III-European Regional Develop. Found); PI22/01684 Bernardino Oliva (Other Grant/Funding Number: Instituto Salud Carlos III-European Regional Develop. Found); PI22/01398 Concepción Violan (Other Grant/Funding Number: Instituto Salud Carlos III-European Regional Develop. Found); PI22/01665 Rafael Rotaeche (Other Grant/Funding Number: Instituto Salud Carlos III-European Regional Develop. Found)
Record Dates: First submitted 2024-06-17; First posted 2024-06-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Multimorbidity
Keywords: Multimorbidity; Primary Health Care; Trajectories; Mixed-methods; Patterns; Qualitative study; Discussion group; Semi-structured interviews; Photovoice; Shared decision-making; Cluster
MeSH Terms: interventions — Retrospective Studies; Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Quantitative Aim: Ambispective longitudinal observational study
  Interventions: Other: Retrospective and prospective cohort
- Qualitative Aim: Focus group, semi-structured interviews and Photovoice
  Interventions: Other: Focus group, semi-structured interviews and Photovoice
- Systematic Review Aim: Systematic literature review on the effectiveness of interventions on training, multimorbidity and polypharmacy in health professionals.
  Interventions: Other: Systematic review

INTERVENTIONS:
Other: Retrospective and prospective cohort — * Retrospective study: Population-based retrospective cohort study with RWD. Patients ≥60 years old with 2 or more chronic diseases diagnosed before 01/01/2012, users of the public health system of the participating Autonomous Communities, will be included. Those who have had no contact with primary care defined as contact in a medical or nursing consultation in the previous two years (2010-2012) will be excluded.
  * Prospective longitudinal observational open cohort study developed in the context of the MULTIPAP and LOXO studies.Patients over 65 years of age with multimorbidity (3 or more chronic pathologies) and polypharmacy (5 or more drugs taken during at least the last 3 months before inclusion in the study) under follow-up from primary care in Madrid, Aragon and Andalusia.
  Groups: Quantitative Aim
Other: Focus group, semi-structured interviews and Photovoice — The participants will be people with multimorbidity over 60 years of age recruited from Primary Care centers in Spain. A theoretical sampling will be carried out. Data will be collected through video and audio recordings from a total of 16 focus groups and 20 interviews in 7 regions, and will finally be transcribed for a triangulated thematic analysis. Two groups will be carried out with participation-action research methodology - Photovoice.
  Groups: Qualitative Aim
Other: Systematic review — No patient recruitment required
  Groups: Systematic Review Aim

SUMMARY:
The overall objective of the study is to analyze the evolution of multimorbidity, its most relevant patterns and trajectories in the Spanish National Health System population, from 2012 to 2022, and to analyze the factors that determine it, as well as the experience of professionals and patients in navigating the health system and in shared decision making.

Multimorbidity trajectories can help identify homogeneous groups of individuals with similar needs and prognoses, and help practitioners and health systems to personalize clinical interventions and preventive strategies. Capturing this dynamism is the only way to better understand the natural history of multimorbidity and shed light on hitherto unexplained findings.

DETAILED DESCRIPTION:
* Design: Mixed-method study.

  * Quantitative study: retrospective and prospective observational study. It integrates demographic and clinical information from electronic medical records and clinical-administrative databases. It involves the harmonisation of the cohorts of users of the public health system of the 7 participating regions.
  * Qualitative study with a phenomenological and ethnographic approach using focus group techniques, semi-structured interviews and Photovoice to find out the perspective of patients and professionals in shared decision-making.
  * Systematic literature review on the effectiveness of interventions on training, multimorbidity and polypharmacy in health professionals.
* Analysis:

  * Quantitative study: Cluster, network and trajectory analysis
  * Qualitative study: Thematic content analysis that will be triangulated among the members of the research team. Meanings will be interpreted and an explanatory framework will be created with the contributions of each type of informant.

ELIGIBILITY:
Inclusion criteria:

* 60 years or older
* 2 or more chronic diseases

Exclusion criteria:

- Not having used the national health system in the last year

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patientes aged 60 years or older with 2 or more chronic diseases diagnosed before 2012-01-01. Population registered at Primary Health Centres in Spain.
  Sampling Method: Not Applicable
Sampling Method: Non-Probability Sample
Enrollment: 3239950 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Multimorbidity | Baseline
  Presence of two or more diagnoses of any of the 60 diseases categorised by the Swedish National Study of Ageing and Care (SNAC-K20) (It is a classification, not a scale)
Death | Start date 31/12/2012, 1 year
  Death and abandonment: the occurrence of this event will be measured, regardless of the cause
Drugs | 1 year
  300 ATC Swedish National Study of Ageing and Care (SNAC-K20) 8It is a classification, not a scale)
Use of service | 1 year
  Primary Care medical/nursing visits, emergencies, referrals, admissions
Morbidity | Baseline/ 1 year
  Defined with ICD-10, laboratory defined in the Swedish National Study of Ageing and Care (SNAC-K20). It is a classification, not a scale
Frailty | Baseline/ 1 year
  EFRAIL (It consists of 5 dichotomous questions. Scoring from 0 to 5. Interpretation:
  * Probable frailty: 3 to 5 points.
  * Probable pre-fragility: 1 to 2 points.
  * No fragility or robustness: 0 points)

SECONDARY OUTCOMES:
Adherence | Baseline
  Morisky-Green (Patients who answer NO to all four questions are considered compliant with treatment and those who answer YES to one or more are considered non-compliant)
Social support | Baseline
  Dukes-Unk-11(This questionnaire consists of 11 items and a Likert-type response scale. The score range is between 11 and 55 points. A score equal to or greater than 32 indicates normal support, while a score of less than 32 indicates low perceived social support)
Functioning and disability | Baseline/ 1 year
  WHODAS (It is composed of 36 items that evaluate the following 6 dimensions. The overall score runs a scale from 0 to 100, with higher values indicating greater disability)
Health releated quality of life | Baseline
  Euroqol 5D-5L (It consists of 2 parts - The EQ-5D descriptive system and the Visual Analog Scale (VAS).
  Scale (VAS). In the VAS the individual scores his or her health between two extremes, 0 and 100, the worst and the best state of health imaginable. imaginable)

OTHER OUTCOMES:
Age | Baseline
  Years
Sex | Baseline
  Male/Female
Country | Baseline
  Country of origin
Deprivation Index | Baseline
  MEDEA (Values from 1 to 5. Higher values indicate a more unfavorable socioeconomic situation)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel del Cura González, PhD,MD, Study Director — Gerencia Asistencial de Atención Primaria
Locations (1):
- Isabel del Cura González, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided